CLINICAL TRIAL: NCT02582476
Title: A Randomised, Double-blind, Placebo-controlled, Phase II Clinical Trial With a Cross-over Design Assessing Efficacy of a Single Dose of Bumetanide in Reducing Focal Attack Severity in Hypokalaemic Periodic Paralysis Assessed Using the McManis Protocol
Brief Title: Bumetanide in Hypokalaemic Periodic Paralysis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrolment and end of funding
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 120542
Record Dates: First submitted 2015-08-11; First posted 2015-10-21 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Hypokalemic Periodic Paralysis
Keywords: Hypokalemic Periodic Paralysis; Bumetanide; Periodic Paralysis
MeSH Terms: conditions — Hypokalemic Periodic Paralysis | interventions — Bumetanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bumetanide — Participants will be randomly assigned to either bumetanide or placebo for the first visit. The assigned treatment will be taken by mouth at the onset of a focal attack defined as 40% decrement in ADM CMAP amplitude compared to the maximum CMAP amplitude recorded during or after the exercise. The second assessment will follow an identical protocol to the first, but with the other treatment administered.
Drug: Placebo — Participants will be randomly assigned to either bumetanide or placebo for the first visit. The assigned treatment will be taken by mouth at the onset of a focal attack defined as 40% decrement in ADM CMAP amplitude compared to the maximum CMAP amplitude recorded during or after the exercise. The second assessment will follow an identical protocol to the first, but with the other treatment administered.

SUMMARY:
This is a randomised, double-blind, placebo-controlled phase II clinical trial with a cross-over design to investigate the efficacy of bumetanide in patients with hypokalemic periodic paralysis (HypoPP).

The aim is to assess the efficacy of bumetanide in reducing severity and duration of a focal attack of weakness in a hand muscle.

Twelve participants will be recruited.

DETAILED DESCRIPTION:
Interested patients who provisionally meet inclusion/exclusion criteria will attend NHNN for a screening visit to check study eligibility and to have any questions relating to study participation answered. Each patient will undertake two assessment visits at approximately four weeks apart. Study participants will withhold carbonic anhydrase inhibitor medications for 72 hours prior to assessment visits as is standard for McManis testing and restart their routine treatment immediately after each visit. Participants will be admitted as an NHNN day case. Following baseline assessments a localised attack of weakness will be induced by isometric exercise of the abductor digit minimi (ADM) in the hand as per McManis protocol below. Participants will be randomly assigned to either bumetanide or placebo for the first visit. Identical appearing capsules will be prepared to blind both researcher and participant to treatment allocation. The assigned treatment will be taken by mouth at the onset of a focal attack defined as 40% decrement in ADM CMAP amplitude compared to the maximum CMAP amplitude recorded during or after the exercise. During the admission each patient will be monitored according to the research protocol. At the end of the assessment protocol the participant will be discharged home. The duration of each admission will be approximately 6 hours The second assessment will follow an identical protocol to the first, but with the other treatment administered.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age;
* Diagnosis of genetically confirmed HypoPP;
* Clinical symptoms or signs of active symptomatic disease (at least 1 attack in last 12 months);
* Practising an acceptable method of birth control for the duration of the trial. This will be addressed on Patient Information Sheet for men and women (section 11.4.5);

Exclusion Criteria:

* Inability or unwillingness to provide informed consent;
* People older than 64 years old;
* Other conditions causing hand weakness which could interfere with study measurements (e.g. due to a stroke, trauma or arthritis)
* Patients with a history of cardiac disease, renal failure or moderate to severe hepatic disease. Note: abnormalities in serum transaminases are common in people with HypoPP as they arise from skeletal muscle rather than any specific liver abnormality. Consequently, raised serum bilirubin >20% above the baseline value will be used to identify abnormal liver function;
* Women who are pregnant or breast-feeding;
* Patients with a current or previous history of diabetes, porphyria, symptomatic hypotension, prostatic hypertrophy or difficulty with micturition, allergy to sulfonamides or thiazides;
* Patients on lithium, digoxin, nephro- or ototoxic drugs;
* Patients known to be allergic bumetanide or its excipients;
* Patients with a history of inadequately treated Addison's disease;
* Patients participating in another interventional trial in the previous 1 month.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Focal attack severity one hour after treatment | The effect of treatment on focal attack severity one hour after treatment
  This will be measured as CMAP amplitude expressed as a percent of peak CMAP during or after the McManis exercise.

SECONDARY OUTCOMES:
Focal attack duration | 4 hours
  This will be measured as the time between treatment administration until CMAP returns to 65% of peak CMAP within 4 hours following the treatment intake.
The initial effect of treatment on severity of a focal attack | The initial effect of treatment on severity of a focal attack within the first two hours post treatment
  The effect of treatment on severity of a focal attack within the first two hours (0-2). This will be measured as CMAP amplitude (in percent compared to peak) area under the curve (AUC) from treatment administration until two hours post-treatment.
The late effect of treatment on severity of a focal attack | The late effect of treatment on severity of a focal attack two to four hours post treatment
  The effect of treatment on severity of a focal attack within the last 2 hours (3-4). This will be measured as CMAP amplitude (in percent) AUC from treatment administration during the third and the fourth hours post-treatment.
Safety of Bumetanide assessed by vital signs, physical exam, potassium levels and self-reported adverse events | Safety of Bumetanide in HypoPP within 7 days of each study visit
  Baseline instantaneous potassium measurements as well as laboratory measurements, vital signs (blood pressure/heart rate) and a physical exam including MRC score are done prior to exercise and IMP intake. During the first 4 hours following IMP intake vital signs (blood pressure/heart rate) and instantaneous serum potassium levels are measured frequently as per protocol. Any reported symptoms or adverse events are recorded. In addition intermittent electrophysiological recordings are taken from the non-exercised hand in order to identify the development of a major attack of paralysis early. At the end of the observation period (4 hours after IMP intake) serum potassium levels are measured by the local hospital laboratory and a physical exam is performed including an MRC score. Safety is also assessed by phone call evaluating adverse events reported by the participants and recorded in a diary occurring within 1 week following each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Doreen Fialho, MD, PhD, Principal Investigator — University College London Hospitals
Locations (1):
- MRC Centre for Neuromuscular Disorders, London, United Kingdom

REFERENCES:
- [Background] Wu F, Mi W, Cannon SC. Beneficial effects of bumetanide in a CaV1.1-R528H mouse model of hypokalaemic periodic paralysis. Brain. 2013 Dec;136(Pt 12):3766-74. doi: 10.1093/brain/awt280. Epub 2013 Oct 18. PMID 24142145
- [Background] Wu F, Mi W, Cannon SC. Bumetanide prevents transient decreases in muscle force in murine hypokalemic periodic paralysis. Neurology. 2013 Mar 19;80(12):1110-6. doi: 10.1212/WNL.0b013e3182886a0e. Epub 2013 Feb 20. PMID 23427324
- See also: Queen Square Trial — http://www.cnmd.ac.uk/research/clinical_trial/Bumetanide_clinical_trial